CLINICAL TRIAL: NCT04668599
Title: Cardio-pulmonary Rehabilitation and Its Impact on Sleep Quality; a Prospective Analysis
Brief Title: Cardio-pulmonary Rehabilitation and Sleep Quality
Status: Completed | Type: Observational
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, Vidya Krishnan, Professor, Case Western Reserve University., MetroHealth Medical Center
Other Study IDs: IRB19-00906
Record Dates: First submitted 2020-10-07; First posted 2020-12-16 (Actual); Results first posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Obstructive Pulmonary Disease; Cardiomyopathies; Heart Failure; Restrictive Lung Disease
MeSH Terms: conditions — Lung Diseases, Obstructive; Cardiomyopathies; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with chronic lung or cardiac diseases: This study will focus on patients with obstructive or restrictive lung diseases eligible for pulmonary rehabilitation.
  Patient with cardiac disease such as heart failure, coronary artery disease or cardiomyopathies who are eligible for cardiac rehabilitation will also be included.
  Interventions: Other: Cardiopulmonary rehabilitation

INTERVENTIONS:
Other: Cardiopulmonary rehabilitation — Patients will undergo standardized cardio-pulmonary rehabilitation program.

SUMMARY:
In this prospective cohort study the investigators aim to evaluate the effect of pulmonary rehabilitation on sleep quality. Disturbed sleep is associated with, frequent exacerbations, increase in the severity of disease and increased mortality in chronic obstructive pulmonary disease (COPD). Sleep quality is a good predictor of quality of life in patients with stable COPD. However, there has been little investigation into non-pharmacological methods to improve sleep quality in patients with COPD and heart failure. It is also uncertain, how long the beneficial effects of cardio-pulmonary rehabilitation on sleep quality, if any, usually last. Due to lack of robust data, the investigators sought to find the effect of cardio-pulmonary rehabilitation on sleep quality.

DETAILED DESCRIPTION:
Sleep disorders including poor quality of sleep are common in patients with heart failure, chronic obstructive pulmonary disease (COPD) and, possibly, other chronic lung disorders. These patients complain of difficulty sleeping and sleep fragmentation, often related to symptoms such as cough, sputum production or shortness of breath. Patients with COPD and heart failure commonly have other abnormalities such as nocturnal oxygen desaturation that may further worsen sleep disturbances. Moreover, sleep disordered breathing (SDB), like obstructive sleep apnea syndrome (OSA), has been linked to higher morbidity and mortality if COPD is present (known as Overlap syndrome). In patients with COPD and heart failure, cardio-pulmonary rehabilitation has important health benefits such as improvement in disease related symptoms, exercise tolerance, and health-related quality of life. However, the effect of cardio-pulmonary rehabilitation on sleep quality is controversial. Disturbed sleep is associated with frequent exacerbations, increase in the severity of disease and increased mortality in COPD and heart failure patients.

The investigators hypothesize that cardio-pulmonary rehabilitation results in improved sleep quality in patients with chronic lung disease and heart failure, this may be an important contributor to improved health outcomes after completion of cardio-pulmonary rehabilitation program.

The study will use data from questionnaires filled by the patients before and after completion of cardio-pulmonary rehabilitation. A 3-month follow up survey using the same questionnaires will be conducted to determine the longevity of improved sleep quality (if present). The questionnaires that will be used include Pittsburgh sleep quality index (PSQI), Epworth sleepiness scale (ESS), Berlin questionnaire, COPD assessment test (CAT) for COPD patients, Kansas city cardiomyopathy questionnaire (KCCQ) for heart failure patients, hospital induced anxiety and depression scale (HADS) and insomnia severity index (ISI).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patient who are willing to participate in follow-up survey 3 months after completion of pulmonary rehabilitation.
* Patients who complete rehabilitation for at least 8 weeks.

Exclusion Criteria:

• Not meeting inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Setting: Outpatient
  The study cohort will include patients will chronic lung and heart diseases who meet the inclusion criteria and are to undergo cardiopulmonary rehabilitation in a safety net hospital.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2024-10-11 (Actual); Study Completion 2024-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vidya Krishnan, MD, Principal Investigator — MetroHealth Medical Center
Locations (1):
- Metrohealth medical center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
No current plan to share individual participant data at this time.

REFERENCES:
- [Background] Soler X, Diaz-Piedra C, Ries AL. Pulmonary rehabilitation improves sleep quality in chronic lung disease. COPD. 2013 Apr;10(2):156-63. doi: 10.3109/15412555.2012.729622. Epub 2013 Mar 20. PMID 23514215
- [Background] Omachi TA, Blanc PD, Claman DM, Chen H, Yelin EH, Julian L, Katz PP. Disturbed sleep among COPD patients is longitudinally associated with mortality and adverse COPD outcomes. Sleep Med. 2012 May;13(5):476-83. doi: 10.1016/j.sleep.2011.12.007. Epub 2012 Mar 18. PMID 22429651
- [Background] Scharf SM, Maimon N, Simon-Tuval T, Bernhard-Scharf BJ, Reuveni H, Tarasiuk A. Sleep quality predicts quality of life in chronic obstructive pulmonary disease. Int J Chron Obstruct Pulmon Dis. 2010 Dec 22;6:1-12. doi: 10.2147/COPD.S15666. PMID 21311688
- [Background] Youngstedt SD, O'Connor PJ, Dishman RK. The effects of acute exercise on sleep: a quantitative synthesis. Sleep. 1997 Mar;20(3):203-14. doi: 10.1093/sleep/20.3.203. PMID 9178916
- [Background] McDonnell LM, Hogg L, McDonnell L, White P. Pulmonary rehabilitation and sleep quality: a before and after controlled study of patients with chronic obstructive pulmonary disease. NPJ Prim Care Respir Med. 2014 Jul 10;24:14028. doi: 10.1038/npjpcrm.2014.28. PMID 25010602

RESULTS

PARTICIPANT FLOW:
Groups:
- Patient With Chronic Lung or Cardiac Diseases: This study will focus on patients with obstructive or restrictive lung diseases eligible for pulmonary rehabilitation.
  Patient with cardiac disease such as heart failure, coronary artery disease or cardiomyopathies who are eligible for cardiac rehabilitation will also be included.
  Cardiopulmonary rehabilitation: Patients will undergo standardized cardio-pulmonary rehabilitation program.
Period: Baseline to Completion of Rehab
Arm/Group | Patient With Chronic Lung or Cardiac Diseases
Started | 106
Completed | 63
Not Completed | 43
Period: Completion of Rehab to 3-Month Followup
Arm/Group | Patient With Chronic Lung or Cardiac Diseases
Started | 63
Completed | 63
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patient With Chronic Lung or Cardiac Diseases
Number analyzed (Participants) | 106
Age, Continuous [Mean (Standard Deviation); unit: years] — What scale measures: age, in years, from time of birth to start of pulmonary rehabilitation Scale range: 18 thru 110 (in years) What numbers mean on range: age, in years, from time of birth to start of pulmonary rehabilitation Purpose of the scale: report age of patient (a known risk factor for sleep disordered breathing)
  years | 63 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants] — What scale measures: sex assigned at birth Scale range: Male, Female What numbers mean on range: N/a Purpose of the scale: report sex assigned at birth (a known risk factor for sleep disordered breathing)
  Participants
    Female | 71
    Male | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — What scale measures: ethnicity, as reported by patient Scale range: Hispanic or Latino / not Hispanic or Latino, Unknown or Not Reported What numbers mean on range: N/a Purpose of the scale: report ethnicity to see if it might be a factor that affects the impact of pulmonary rehabilitation on sleep outcomes
  Participants
    Hispanic or Latino | 13
    Not Hispanic or Latino | 93
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — What scale measures: race as reported by patient Scale range: American Indian or Alaska Native, Asian, native Hawaiian or other pacific slander, Black or African American, White, more than one race, Unknown or not reported What numbers mean on range: N/a Purpose of the scale: report race to see if it may be a factor on the association of pulmonary rehabilitation and sleep outcomes
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 35
    White | 71
    More than one race | 0
    Unknown or Not Reported | 0
Body-Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] — What scale measures: body mass index, as measured during first session of pulmonary rehabilitation Scale range: 15 to 100 kg/m2 What numbers mean on range: calculated body mass index based on height and weight.
  Purpose of the scale: report body mass index, a known risk factor for sleep disordered breathing.
  kg/m2 | 29.9 (7.2)
Epworth Sleepiness Scale [Median (Inter-Quartile Range); unit: units on a scale] — What scale measures: reported sleepiness of patient in passive and active scenarios.
  Scale range: 0 through 24 What numbers mean on range: higher numbers indicated more sleepiness. Epworth > 10 is considered pathologically sleepy.
  Purpose of the scale: report patient-reported sleepiness to see if it correlates with any objective measures of sleep outcomes.
  units on a scale | 9 [5 to 11]

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Sleep Quality Using Pittsburgh Sleep Quality Index
Description: Pittsburgh sleep quality index is validated questionnaire and will be used to determine improvement in sleep quality before and after completion of cardiopulmonary rehabilitation. Pittsburgh sleep quality index comprises of seven components. Each component is marked from 0 to 3, with a maximum total score of 21 and a minimum total score of 0. A score of less than 5 indicates good overall sleep quality and a score of 5 and more indicates poor sleep quality.
  From literature review using Pittsburgh sleep quality index, minimal clinically important difference was determined to be 3 between before and after measurements.
Time Frame: 8 weeks on average
Population: those who completed PR (8 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Patients Who Completed Rehab (8 Weeks): This study will focus on patients with obstructive or restrictive lung diseases eligible for pulmonary rehabilitation.
  Patient with cardiac disease such as heart failure, coronary artery disease or cardiomyopathies who are eligible for cardiac rehabilitation will also be included.
  Cardiopulmonary rehabilitation: Patients will undergo standardized cardio-pulmonary rehabilitation program.
- Patients Who Completed Rehab and 3-month Followup (5 Months): patients who completed pulmonary rehabilitation and 3-month followup - this would be the 8 weeks of rehab plus 3 months so 5 months in total
Arm/Group | Patients Who Completed Rehab (8 Weeks) | Patients Who Completed Rehab and 3-month Followup (5 Months)
Number analyzed (Participants) | 63 | 59
units on a scale | -3.6 (2.7) | -1.6 (2.8)

2. Secondary Outcome: Change in Insomnia Severity Index
Description: Insomnia severity index will be determined before and after cardiopulmonary rehabilitation. Insomnia severity index consists of 7 items with a minimum total score of 0 and maximum total score of 28 with a score of 8 or more suggesting presence of insomnia. A 6 point change is considered significant (minimum significant important difference) as determined by literature. Paired student t-test will be used to compare means before and after cardio-pulmonary rehabilitation
Time Frame: 8 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Patients Who Completed Rehab: This study will focus on patients with obstructive or restrictive lung diseases eligible for pulmonary rehabilitation.
  Patient with cardiac disease such as heart failure, coronary artery disease or cardiomyopathies who are eligible for cardiac rehabilitation will also be included.
  Cardiopulmonary rehabilitation: Patients will undergo standardized cardio-pulmonary rehabilitation program.
- Patients Who Completed Followup: Pulm and cardiac rehab patients who completed rehab and the 3 month followup
Arm/Group | Patients Who Completed Rehab | Patients Who Completed Followup
Number analyzed (Participants) | 63 | 58
units on a scale | -5 (2.6) | -2.8 (3.8)

ADVERSE EVENTS:
Time Frame: Eight weeks + 3 months. the eight weeks represents the duration of the pulmonary rehabilitation, and the additional 3 months is the follow-up after pulmonary rehabilitation.
Arm/Group | Patient With Chronic Lung or Cardiac Diseases
All-Cause Mortality (participants affected / at risk) | 0/106
Serious Adverse Events (participants affected / at risk) | 0/106
Other Adverse Events (participants affected / at risk) | 0/106

LIMITATIONS AND CAVEATS:
Rehab moved from main campus to off-site, limiting our ability to recruit more patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-11-05): https://cdn.clinicaltrials.gov/large-docs/99/NCT04668599/Prot_003.pdf
  • Statistical Analysis Plan (2020-05-10): https://cdn.clinicaltrials.gov/large-docs/99/NCT04668599/SAP_000.pdf
  • Informed Consent Form (2020-05-10): https://cdn.clinicaltrials.gov/large-docs/99/NCT04668599/ICF_002.pdf